CLINICAL TRIAL: NCT04062305
Title: Feasibility of Navigated Transcranial Magnetic Stimulation (nTMS) of Patients Treated With Stereotactic Radiosurgery for Brain Metastases in the Motor Cortex: A Comprehensive Cross-Sectional Assessment
Brief Title: nTMS in Planning Stereotactic Radiosurgery in Patients With Brain Metastases in the Motor Cortex
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-0302; NCI-2019-04992 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0302 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Radiation Therapy Recipient
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (nTMS, sensory testing) (Experimental): Patients undergo nTMS over 1 hour. Patients also perform 4 tasks that test grip and pinch strength, and the ability to use and feel with their hands for 1 hour.
  Interventions: Behavioral: Hand Function Test; Procedure: Navigated Transcranial Magnetic Stimulation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Hand Function Test — Complete tasks that test grip strength, pinch strength, and ability to use and feel with hands
  Other Names: Hand Sensory Test
Procedure: Navigated Transcranial Magnetic Stimulation — Undergo nTMS
  Other Names: Navigated TMS; nTMS
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well nTMS works in planning for stereotactic radiosurgery in patients with brain metastases in the motor cortex. Stereotactic radiosurgery is a type of radiation therapy that delivers high doses of radiation, which can sometimes lead to damage occurring to the brain and surrounding areas. The motor cortex (the part of the nervous system that controls muscle movement), however, currently has no radiation dose limit. nTMS is a non-invasive tool that uses sensors on a patient's muscle to trace the location in their brain that controls that muscle and is currently used by doctors to decide where to operate so as not to damage the motor nerves. nTMS may effectively help plan radiation treatment using SRS and help doctors decide on how much radiation can be used on motor nerves.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the use of navigated transcranial magnetic stimulation (nTMS) in the radiation oncology clinic is feasible.

SECONDARY OBJECTIVES:

I. To investigate the relationship of stereotactic radiosurgery (SRS) dosimetry and lesion involvement in the motor tracts identified using nTMS and the presence or absence of motor deficits evaluated by objective and subjective measures (Manual Ability Measure [MAM]-20, Euroqol [EQ]-5 Dimensional [D]-5 Level [L], and MD Anderson Symptom Inventory [MDASI]-Brain Tumor [BT] questionnaires).

II. To determine if nTMS of contralateral motor tracts provides a viable internal control, considering handedness.

III. To aid in the design of a prospective, randomized clinical trial that will limit radiation dose to brain metastases located in close proximity to the motor cortex with the goal of improving functional and quality of life outcomes measured by occupational therapy tasks and the MAM-20, EQ-5D-5L, and MDASI-BT questionnaires.

IV. To explore the utility of electroencephalography (EEG) in correlation with nTMS and reported functional outcomes measured by occupational therapy tasks and the MAM-20, EQ-5D-5L, and MDASI-BT questionnaires.

OUTLINE:

Patients undergo nTMS over 1 hour. Patients also perform 4 tasks that test grip and pinch strength and the ability to use and feel with their hands for 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with brain metastases located in or near the motor cortex who have previously received SRS to that lesion within the prior 3-18 months
* Patients must be able to participate in nTMS of bilateral motor cortices
* Patients must be able to participate in an electromyography (EMG)
* Patient's must have utilized magnetic resonance imaging (MRI) for their previous SRS treatment planning
* Patient must be able to complete the Functional and Quality of Life questionnaires in English

Exclusion Criteria:

* Significant cognitive or psychiatric symptoms that prevent the ability to complete a physical exam, questionnaires, or participate in nTMS or EMG
* Poor performance status Karnofsky performance score (KPS < 60) that prevents the ability to participate in a physical exam, nTMS, or EMG. Patients will not be excluded if they are not able to complete the exploratory EEG analysis
* Patients receiving any prior treatment that might impact their cognitive, psychiatric, or motor cortex function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2027-05-06 (Estimated); Study Completion 2027-05-06 (Estimated)

PRIMARY OUTCOMES:
Operational feasibility of navigated transcranial magnetic stimulation (nTMS) | Up to 1 year
  Will be determined to be operationally feasible on a patient if the images and data obtained from nTMS for the patient provide useful information to the radiation oncologist and if the radiation oncologist determines that this additional information would improve patient care. Will deem the use of nTMS to be operationally feasible overall if it is deemed operationally feasible on an underlying proportion of at least 90% potentially consented patients. Will calculate the proportions of operational and technical feasibility of the use of nTMS and their 80% confidence intervals (CIs). If the observed proportions are greater than or equal to 82%, the use of nTMS to be operationally and technically will be deemed feasible.
Technical feasibility of nTMS | Up to 1 year
  Will be determined to be technically feasible on a patient if the procedure of nTMS is able to be performed on the patient, resulting in mapped motor cortex data. If the patient is not able to complete the procedure for any reason, that patient's nTMS treatment will not be technically feasible. Will deem the use of nTMS to be technically feasible overall if it is deemed technically feasible on an underlying proportion of at least 90% potentially consented patients. Will calculate the proportions of operational and technical feasibility of the use of nTMS and their 80% CIs. If the observed proportions are greater than or equal to 82%, the use of nTMS to be operationally and technically will be deemed feasible.
Economic feasibility of nTMS | Up to 1 year
  Will be determined to be economically feasible if there are no additional costs to the patients and department, other than those outlined in the proposed budget.
Identification of the motor cortex by addition of nTMS | Up to 1 year
  The treating radiation oncologist will determine if the use of nTMS provides additional information over the standard atlas-based definition of the motor region if they state that they would have made adjustments to their treatment volume of the tumor based on the new nTMS data provided.

SECONDARY OUTCOMES:
Stereotactic radiosurgery (SRS) dosimetry and lesion involvement in the motor tracts | Up to 1 year
  The relationship will be identified using nTMS. Dose volume histogram data for the motor cortex and motor tracts will be generated.
Presence or absence of motor deficits | Up to 1 year
  Will be determined by the Manual Ability Measure-20, Euroqol-5 Dimensional-5 Level, and MD Anderson Symptom Inventory - Brain Tumor questionnaires. Data analyses will be performed to determine correlations between objective/subjective deficits (based on the results of the questionnaires) and dose volume histogram data for the motor cortex and tracts.
Production of viable internal control by contralateral motor tract, accounting for handedness | Up to 1 year
Development of a clinical trial that will limit radiation dose to brain metastases | Up to 1 year
  Will determine if trial can aid in the design of a prospective, randomized clinical trial that will limit radiation dose to brain metastases located in close proximity to the motor cortex with the goal of improving functional and quality of life outcomes based on meeting the primary objective of this study.
Utility of electroencephalography (EEG) | Up to 1 year
  The utility of EEG in correlation with nTMS and reported functional outcomes will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Chung, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT04062305/ICF_000.pdf